CLINICAL TRIAL: NCT03318861
Title: A Phase 1 Multicenter Study of KITE-585, an Autologous Anti-BCMA CAR T-Cell Therapy, in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study to Evaluate the Safety and Efficacy of KITE-585 in Participants With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KITE-585-501
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Results first posted 2020-05-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Dose-Escalation and Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation: 3 x 10^7 KITE-585 (Experimental): Participants with relapsed/refractory multiple myeloma (RRMM), will receive conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day intravenous (IV) infusion for 3 days followed by a single infusion of KITE-585 at a dose of 3 x 10^7 autologous anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR) T cells on Day 0. Participants may also receive an optional bridging therapy at the investigator's discretion, up to 7 days before initiation of conditioning chemotherapy. Participants will then have a post-treatment assessment period and long-term follow-up period from Week 2 to Month 3 and after Month 3 to Year 15, respectively.
  Interventions: Genetic: KITE-585; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Escalation: 1 x 10^8 KITE-585 (Experimental): Participants with RRMM, will receive conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 1 x 10^8 autologous anti-BCMA CAR T cells on Day 0. Participants may also receive an optional bridging therapy at the investigator's discretion, up to 7 days before initiation of conditioning chemotherapy. Participants will then have a post-treatment assessment period and long-term follow-up period from Week 2 to Month 3 and after Month 3 to Year 15, respectively.
  Interventions: Genetic: KITE-585; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Escalation: 3 x 10^8 KITE-585 (Experimental): Participants with RRMM, will receive conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 3 x 10^8 autologous anti-BCMA CAR T cells on Day 0. Participants may also receive an optional bridging therapy at the investigator's discretion, up to 7 days before initiation of conditioning chemotherapy. Participants will then have a post-treatment assessment period and long-term follow-up period from Week 2 to Month 3 and after Month 3 to Year 15, respectively.
  Interventions: Genetic: KITE-585; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Escalation: 1 x 10^9 KITE-585 (Experimental): Participants with RRMM, will receive conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 1 x 10^9 autologous anti-BCMA CAR T cells on Day 0. Participants may also receive an optional bridging therapy at the investigator's discretion, up to 7 days before initiation of conditioning chemotherapy. Participants will then have a post-treatment assessment period and long-term follow-up period from Week 2 to Month 3 and after Month 3 to Year 15, respectively.
  Interventions: Genetic: KITE-585; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585 (Experimental): RRMM participants with moderate renal impairment (creatinine clearance 30 to 59 mL/min [Grade 2 chronic kidney disease]) will receive a conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 24 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a tolerable dose of 3 x 10^7 autologous anti-BCMA CAR T cells on Day 0. Participants may also receive an optional bridging therapy at the investigator's discretion, up to 7 days before initiation of conditioning chemotherapy. Participants then had a post-treatment assessment period and long-term follow-up period from Week 2 to Month 3 and after Month 3 to Year 15, respectively.
  Interventions: Genetic: KITE-585; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Genetic: KITE-585 — A single infusion of KITE-585 autologous anti-BCMA CAR T cells
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of KITE-585, an autologous engineered chimeric antigen receptor (CAR) T-cell product targeting a protein commonly found on myeloma cells called B-cell maturation antigen (BCMA), as measured by the incidence of dose-limiting toxicities (DLTs). Participants will be given a 3 day course of conditioning chemotherapy followed by a single infusion of KITE-585.

DETAILED DESCRIPTION:
Participants with relapsed/refractory multiple myeloma can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, ECG and echocardiogram of the heart, brain MRI, and blood draws. Eligible participants have white blood cells collected by leukapheresis. These cells are genetically modified to make the experimental treatment KITE-585. Participants receive conditioning chemotherapy prior to the KITE-585 infusion. After the KITE-585 infusion, participants will be followed for side effects and effect of KITE-585 on their myeloma. Study procedures may be performed while hospitalized and/or in the outpatient setting. Participants who received an infusion of KITE-585 will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Key Inclusion Criteria:

1. Measurable relapsed or refractory myeloma as defined by the International Myeloma Working Group (IMWG) Consensus Criteria following treatment with at least 3 lines of therapy including with both a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD), or progressive myeloma that is refractory to a regimen containing both a PI and an IMiD.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Adequate bone marrow, renal, hepatic, pulmonary, and cardiac function defined as:

   * Absolute neutrophil count (ANC) ≥ 1,000/µL
   * Platelet count ≥ 75,000/µL
   * Absolute lymphocyte count ≥ 100/µL
   * Creatinine clearance above limits set in the protocol for each cohort
   * Normal cardiac function as assessed by electrocardiogram (ECG) and echocardiogram
   * Baseline oxygen saturation > 92% on room air and no clinically significant pleural effusion

Key Exclusion Criteria:

1. Plasma cell leukemia
2. Non-secretory multiple myeloma
3. History of Central nervous system (CNS) involvement by multiple myeloma
4. Prior CAR therapy or other genetically modified T cells
5. Inadequate washout from prior therapy
6. Autologous stem cell transplant within 6 weeks before enrollment or any history of allogenic transplant
7. History of active autoimmune disease
8. History of deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months before enrollment
9. Recent history of other (non multiple myeloma) cancer
10. Active viral, fungal, bacterial or other infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (9):
- United States (9):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornell RF, Bishop MR, Kumar S, Giralt SA, Nooka AK, Larson SM, Locke FL, Raje NS, Lei L, Dong J, Le Gall JB, Rossi JM, Orlowski RZ. A phase 1, multicenter study evaluating the safety and efficacy of KITE-585, an autologous anti-BCMA CAR T-cell therapy, in patients with relapsed/refractory multiple myeloma. Am J Cancer Res. 2021 Jun 15;11(6):3285-3293. eCollection 2021. PMID 34249462
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KITE-585-501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 21 participants were screened.
Groups:
- Dose Escalation: 3 x 10^7 KITE-585: Participants with relapsed/refractory multiple myeloma (RRMM), received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day intravenous (IV) infusion for 3 days followed by a single infusion of KITE-585 at a dose of 3 x 10^7 autologous anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR) T cells on Day 0.
- Dose Escalation: 1 x 10^8 KITE-585: Participants with RRMM, received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 1 x 10^8 autologous anti-BCMA CAR T cells on Day 0.
- Dose Escalation: 3 x 10^8 KITE-585: Participants with RRMM, received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 3 x 10^8 autologous anti-BCMA CAR T cells on Day 0.
- Dose Escalation: 1 x 10^9 KITE-585: Participants with RRMM, received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 1 x 10^9 autologous anti-BCMA CAR T cells on Day 0.
- Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585: RRMM participants with moderate renal impairment (creatinine clearance 30 to 59 mL/min [Grade 2 chronic kidney disease]) received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 24 mg/m^2/day IV infusion for 3 days followed by single infusion of KITE-585 at a tolerable dose of 3 x 10^7 autologous anti-BCMA CAR T cells on Day 0.
Period: Overall Study
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Started | 3 | 4 | 3 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 4 | 3
Not completed — Death | 2 | 3 | 3 | 2 | 2
Not completed — Enrolled But Never Treated | 0 | 1 | 0 | 1 | 1
Not completed — Informed Consent Withdraw | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal of Consent From Further Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who were enrolled in the study.
Groups:
- Dose Escalation: 3 x 10^7 KITE-585: Participants with RRMM, received conditioning chemotherapy consisting of cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day IV infusion for 3 days followed by a single infusion of KITE-585 at a dose of 3 x 10^7 autologous anti-BCMA CAR T cells on Day 0.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 4 | 2 | 14
  >=65 years | 0 | 1 | 1 | 0 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.3 [50 to 56] | 59.8 [49 to 71] | 59.3 [49 to 67] | 54.3 [47 to 58] | 56.3 [47 to 65] | 56.5 [47 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 2 | 7
  Male | 3 | 3 | 1 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 3 | 4 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 1 | 3 | 3 | 13
  Black or African American | 0 | 1 | 1 | 1 | 0 | 3
  Other | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: A DLT is a KITE-585-related event with onset in the first 28 days following infusion. DLTs are defined by events and duration of events, including:
  * Any duration: Grade (GR) 4 cytokine release syndrome (CRS), KITE-585-related GR 5 adverse events (AE) and GR 4 nonhematologic AE with the exceptions of fever, nausea, hepatic toxicity that resolves to GR 3 or better in ≤ 72 hours, hypogammaglobulinemia, tumor lysis syndrome, acute renal toxicity requiring dialysis for ≤ 7 days, intubation for airway protection for ≤ 7 days and AE resolves to ≤ GR 1 within 2 weeks and baseline within 4 weeks
  * ≥ 72 hours: GR 3 CRS and GR 3 nonhematologic AE with the exceptions of fever, nausea, hepatic toxicity that resolves to GR 2 or better in ≤ 14 days, hypogammaglobulinemia and tumor lysis syndrome
  * ≥ 30 days: GR 4 hematologic AE with the exceptions of cytopenias attributable to ongoing or recurrent multiple myeloma
Time Frame: From KITE-585 infusion until 28 days after KITE-585 infusion
Population: DLT Evaluable Set included participants in the dose escalation period who received the target dose (± 20%) and were followed for at least 28 days after the first KITE-585 infusion; or received a dose of KITE-585 lower than 20% below the target dose for that cohort and experienced a DLT during the 28-day post-first-infusion period.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585
Number analyzed (Participants) | 3 | 4 | 3 | 4
percentage of participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR) as Determined by Study Investigators According to the International Myeloma Working Group (IMWG) Consensus Panel 1 Criteria
Description: ORR: Percentage of participants who achieved a stringent CR (sCR), complete response (CR), partial response (PR), or very good PR (VGPR), as determined by IMWG Consensus Panel 1 Criteria. sCR: CR+normal free light chain (FLC) ratio, no clonal cells in BM by immunohistochemistry or immunofluorescence; CR: negative immunofixation (IFX) on serum and urine, no soft tissue plasmacytomas (STP), <5% plasma cells in bone marrow (BM); PR: ≥50% decrease of serum M-protein + 24hr urinary M-protein decrease by ≥90% or <200 mg/24hr. If unmeasurable serum and urine M-protein; and serum-free light assay; requires ≥ 50% decrease in the difference between involved and uninvolved FLC levels / ≥ 50% reduction in plasma cells (PC), provided baseline BM PC percentage was ≥ 30%, respectively. If present at baseline, ≥ 50% reduction in the size of STP is also required; VGPR: serum and urine M-protein detected by IFX but not electrophoresis, >90% in serum M-protein+urine, M-protein level <100 mg/24hr.
Time Frame: From KITE-585 infusion to the earlier date of data cutoff and first administration of other anti-cancer therapies including stem cell transplant (maximum: 17.6 months)
Population: The Safety Analysis Set included all participants treated with any dose of KITE-585.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
percentage of participants | 33.3 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS) as Determined by Study Investigators According to the IMWG Consensus Panel 1
Description: PFS: Interval from first study drug dose date to the earlier of first documentation of definitive progressive disease (PD) per IMWG Consensus Panel 1 Criteria or death from any cause. PD: an increase of 25% from the lowest response value in 1 of the following: Serum and urine M-protein (absolute increase ≥ 0.5 g/dL and ≥ 200 mg/24 hours, respectively); In participants without measurable serum and urine M-protein levels, the difference between involved and uninvolved FLC levels (absolute increase > 10 mg/dL); In participants without measurable serum and urine M-protein and without measurable disease by FLC levels, bone marrow PC percentage (absolute percentage ≥ 10%). Definite development of new bone lesions or STP or definite increase in the size of existing bone lesions or STPs; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder. Analysis was done using Kaplan-Meier (KM) estimate.
Time Frame: as for outcome 2
Population: Participants in the Safety Analysis Set were analyzed. Participants not meeting the criteria for PD by the analysis data cutoff date were censored at their last evaluable disease assessment date before any other anti-cancer therapies including stem cell transplant.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
months | 1.1 [0.5 to 3.2] | 1.0 [0.9 to 1.0] | 0.8 [0.5 to 1.0] | 1.0 [0.9 to 1.0] | NA [2.0 to NA] — Median and upper limit of confidence interval (CI) were not estimable due to insufficient number of events.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first dose date of study drug to the date of death from any cause. Analysis was done using KM estimate. Participants who have not died by the analysis data cutoff date were censored at their last date known to be alive or cutoff date, whichever is earlier.
Time Frame: From KITE-585 infusion to date of data cutoff (maximum: 17.6 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
months | NA [11.1 to NA] — Median and upper limit of CI were not estimable due to insufficient number of events. | 5.1 [3.0 to NA] — Upper limit of CI was not estimable due to insufficient number of events. | 6.9 [3.2 to NA] — Upper limit of CI was not estimable due to insufficient number of events. | NA [5.5 to NA] — Median and upper limit of CI were not estimable due to insufficient number of events. | 12.2 [NA to NA] — Lower and upper limit of CI were not estimable due to insufficient number of events.

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: Enrollment through 24 months after treatment with KITE-585 or up to disease progression or initiation of another anti-cancer therapy, whichever occurs first (maximum: 2.9 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities
Description: Clinically significant laboratory abnormalities were defined as per investigator's discretion.
Time Frame: as for outcome 5
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Duration of Response (DOR) as Determined by Study Investigators According to the IMWG Consensus Panel 1
Description: DOR is defined for participants who experience an objective response and is defined as the time from the date of their first objective response (which is subsequently confirmed) to PD per IMWG Consensus Panel 1 Criteria or death from any cause, whichever is earlier. Objective response is defined in Outcome measure 2.
Time Frame: From first response to the earlier date of data cutoff and first administration of other anti-cancer therapies including stem cell transplant (maximum: 17.6 months)
Population: Participants in the Safety Analysis Set who achieved a stringent CR (sCR), complete response (CR), partial response (PR), or very good PR (VGPR), as determined by IMWG Consensus Panel 1 Criteria were to be analyzed. As per changes in planned analysis, this outcome measure could not be analyzed at the data cutoff date due to an insufficient number of responders. Kite/Gilead did not collect the DOR data after the data cutoff date.
Measure: Number; unit: months
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
months | NA — Due to an insufficient number of responders, this endpoint was not analyzed. |  |  |  |

8. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT is defined as the length of time between the date of KITE-585 infusion to the date of initiation of the next therapy or death due to any cause, whichever is earlier.
Time Frame: as for outcome 2
Population: Participants in the Safety Analysis Set were to be analyzed. Estimates of the proportion of participants who have not required additional treatment for progressive multiple myeloma at selected time points were to be provided. As per changes in planned analysis, this outcome measure could not be analyzed at the data cutoff date due to a lack of events. Kite/Gilead did not collect data to analyze TTNT after the data cutoff date.
Measure: Number; unit: months
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
months | NA — Due to lack of events, this outcome measure was not analyzed. | NA — Due to lack of events, this outcome measure was not analyzed. | NA — Due to lack of events, this outcome measure was not analyzed. | NA — Due to lack of events, this outcome measure was not analyzed. | NA — Due to lack of events, this outcome measure was not analyzed.

ADVERSE EVENTS:
Time Frame: Adverse Events: Enrollment through 24 months after treatment with KITE-585 or up to disease progression or initiation of another anti-cancer therapy, whichever occurs first. (maximum: 2.9 months) All-Cause Mortality: Enrollment up to 57.6 months
Description: Adverse Events: The Safety Analysis Set included all participants treated with any dose of KITE-585.
  All-Cause Mortality: The Full Analysis Set included all participants who were enrolled in the study.
Arm/Group | Dose Escalation: 3 x 10^7 KITE-585 | Dose Escalation: 1 x 10^8 KITE-585 | Dose Escalation: 3 x 10^8 KITE-585 | Dose Escalation: 1 x 10^9 KITE-585 | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/4 | 3/3 | 3/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 3 x 10^7 KITE-585 (N=3) | Dose Escalation: 1 x 10^8 KITE-585 (N=3) | Dose Escalation: 3 x 10^8 KITE-585 (N=3) | Dose Escalation: 1 x 10^9 KITE-585 (N=3) | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585 (N=2)
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: 3 x 10^7 KITE-585 (N=3) | Dose Escalation: 1 x 10^8 KITE-585 (N=3) | Dose Escalation: 3 x 10^8 KITE-585 (N=3) | Dose Escalation: 1 x 10^9 KITE-585 (N=3) | Dose Expansion (Renal Impairment): 3 x 10^7 KITE-585 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 1 | 3 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Thyroxine decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 2 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 2
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Amendment 2 (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03318861/Prot_000.pdf
  • Study Protocol: Amendment 3 (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03318861/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03318861/SAP_001.pdf